CLINICAL TRIAL: NCT03468842
Title: Randomized, Double-blind, Placebo-controlled Parallel Group Study to Evaluate the Clinical Efficacy of Streptococcus Dentisani CECT 7746 in Caries Risk Reduction
Brief Title: Study to Evaluate the Clinical Efficacy of Streptococcus Dentisani CECT 7746 in Caries Risk Reduction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AB Biotics, SA (Industry)
Collaborators: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABB-DENTISANI-2015
Record Dates: First submitted 2018-02-26; First posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-02

CONDITIONS: Caries
Keywords: Streptococcus dentisani; caries; salivary pH; S. mutans
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: The study will follow a randomized, double-blind, placebo-controlled design with 2 parallel prospective follow-up groups.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Composition: excipients without probiotic: 2%w/v Guam guar and 6% w/v hydroxyethilcellulose Application in mouth of a bucoadhesive gel. Applied by the profesional at days 0, 15 and 30 and by the participants the rest of the days Frequency: each 48 h by the participants Duration: during 30 days
  Interventions: Biological: Placebo
- Probiotic (Active Comparator): Composition: Streptococcus dentisani: 2,5E+09CFUs, 2% (p/v) Guam Guar and 6% (p/v) Hidroxietilcelulosa. Dose of 2.5E+09 cfu/vial considering one administration every 48 hours, it will be equivalent to a dose of 1.0E+10 cfu/week Application in mouth of a bucoadhesive gel. Applied by the profesional at days 0, 15 and 30 and by the participants the rest of the days Frequency: each 48 h by the participants Duration: during 30 days
  Interventions: Biological: Probiotic

INTERVENTIONS:
Biological: Probiotic — Already described
  Arms: Probiotic
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Exploratory, phase I study to evaluate the clinical efficacy of Streptococcus dentisani CECT 7746 in the risk reduction of caries. Patients who meet the inclusion and exclusion criteria will be randomized and receive the corresponding treatment. The study will follow a randomized design, with two groups in parallel (placebo group and probiotic group) of prospective, double-blind follow-up, for a period of 45 days. The present study will be conducted in a single center and will include a total of 70 patients. The present study has a double main objective:

* Evaluate whether the administration of the probiotic S. dentisani CECT 7746 alkalizes the basal pH of saliva.
* Test the safety and tolerability of the probiotic

Secondary

* Evaluate other microbiological parameters associated with caries risk such as the presence of microorganisms such as S. mutans.
* Evaluate the presence in the mouth and colonization capacity of S. dentisani.
* Evaluate the lactic acid and the pH of the ex vivo plate before and after the administration of a sugar solution
* Evaluate the salivary pH before and after the administration of a sugar solution
* Evaluate the salivary pH before brushing with water.
* Evaluate the buffer capacity of saliva

DETAILED DESCRIPTION:
The probiotic Streptococcus dentisani is a bacterial species present in the human oral microbial flora. It was isolated initially, as result of observation and hypothesis, of volunteers who had never developed caries. These strains have demonstrated, through in vitro studies, an enormous potential of inhibition against S. mutans, besides inhibiting the growth of other pathogens commonly present in common oral pathologies (gingivitis, periodontitis or halitosis). The probiotic product has been shown to be effective in in vitro experiments, artificial mouth models and epidemiological data, statistically significant. However, it is necessary to document the efficacy of Streptococcus dentisani in an oral application study.

Recruitment visit:

In a first visit, it will be assessed if the candidates meet all the inclusion criteria and none of the exclusion criteria. For this, a dental revision will be carried out to assess the different parameters (plaque index, gingival index and salivary flow among others), and a saliva sample will be taken after brushing with water to determine its basal pH.

Those participants who meet the criteria and provide written informed consent will be assigned to one of the two treatment groups (probiotic or placebo). The assignment will be done randomly using a computer generated list.

In this first visit, an impression of the jaw will also be made of those volunteers who meet the criteria and have been randomized. This impression will be used to manufacture custom splints that allow a more comfortable application of the treatment during the study by the participants.

A detailed list of probiotic products present in the market for oral use will be provided.

Basal visit (Day 0):

After 1-2 weeks of the recruitment visit, participants will return to the center for the baseline visit. During this visit, samples of saliva (2 ml) and plaque (from quadrants 1 and 3 on the vestibular and lingual surfaces) will be taken for the quantification and detection of S. mutans and Streptococcus dentisani, and plaque samples of quadrants 2 and 4 by the vestibular and lingual surfaces to quantify the lactic acid produced by the ex vivo plaque, and its pH. The pH of the saliva will also be evaluated before and after brushing with only water and then measured before and after a rinse with active movements with 10 ml of a 10% sugar solution for 1 minute. Finally, the buffering capacity of the saliva, measured by the amount of acid that the saliva is capable of buffering using reactive strips, will be evaluated.

The participants will be treated with probiotic or placebo, depending on the group to which they have been assigned, without the participant or the researcher knowing the assigned treatment. For this the two products will present the same appearance. The randomization will remain blind until the end of the study.

The treatment will consist of the application of the product in the form of gel by all the free surfaces of the teeth by means of a splint. The production of the splints will be done by the same recruiting center. These are washable and reusable splints during the entire study treatment.

The first treatment will be carried out during the baseline visit and will be applied by the clinic professional, who will explain to the participant how to perform successive applications at home every 48 hours.

Participants will receive the splint and the exact number of doses of probiotic or placebo needed for the next visit, which they should return in a bag to verify that the treatment has been followed correctly. Likewise, volunteers will receive a fluoride toothpaste (1000 ppm), a toothbrush and instructions on how to maintain healthy hygiene habits to standardize study conditions. The use of mouthwashes and oral probiotic consumption will be expressly prohibited during the study, all participants will receive a copy of Annexes I and II with the list of mouthwash and probiotic products not admitted.

Visit 1 (Day 15 ± 2 days, follow-up visit):

In this visit participants will be asked to deliver the unused material and they will be provided with the treatments in the exact dosage number until the next visit, as well as the elements for oral hygiene. The appearance of any adverse effect during the consumption of the product will be reviewed with the patient, for it a dental revision will be carried out to evaluate different parameters (plaque index, gingival index and salivary flow among others). During this visit, samples of saliva (2 ml) and plaque (from quadrants 1 and 3 on the vestibular and lingual surfaces) will be taken for the quantification and detection of S. mutans and Streptococcus dentisani, and plaque samples of quadrants 2 and 4 by the vestibular and lingual surfaces to quantify the lactic acid produced by the ex vivo plaque, and its pH. The pH of the saliva will also be evaluated before and after brushing with only water and then measured before and after a rinse with active movements with 10 ml of a 10% sugar solution for 1 minute. Finally, the buffer capacity of saliva will be evaluated.

During this visit, the clinic professional will once again apply the product to all participants and remind them how successive applications should be made at their home every 48 hours.

Visit 2 (Day 30 ± 2 days, end of treatment):

The same procedure will be followed as in visit 1 (day 15), but new single doses will not be provided.

Visit 3 (Day 45 ± 2 days, final visit):

During this visit, samples of saliva (2 ml) and plaque (from quadrants 1 and 3 on the vestibular and lingual surfaces) will be taken for the quantification and detection of S. mutans and Streptococcus dentisani, and plaque samples of quadrants 2 and 4 by the vestibular and lingual surfaces to quantify the lactic acid produced by the ex vivo plaque, and its pH. The pH of the saliva will also be evaluated before and after brushing with only water and then measured before and after a rinse with active movements with 10 ml of a 10% sugar solution for 1 minute. Finally, the buffer capacity of saliva will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 and 65
* With a previous history of caries and / or active cavities
* Absence of other oral diseases
* With a basal oral pH (after brushing with only water) in saliva equal to or less than 7

Exclusion Criteria:

* Antibiotic use during the 30 days prior to the start of the study.
* Usual consumption of chlorhexidine or other mouthwashes with bactericidal active ingredients during the 30 days prior to the start of the study.
* Consumption of oral probiotics during the 30 days prior to the start of the study (Annex II)
* Pregnant or lactating women
* Participants with chronic diseases (eg diabetes, kidney problems, cancer) or who may affect the salivary flow
* Participants in chronic treatment or with medication that can reduce salivary flow, such as antidepressants or psychotropic drugs.
* Allergy to any of the ingredients of the research product

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-05-13 (Actual); Primary Completion 2017-03-24 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline Salivary pH before and after brushing with wáter at 15, 30 and 45 days | Through study completion, an average of 9 months
  Increase in salivary pH measured on the RQflex 10 reflectometer using Reflectoquant test strips at 15, 30 and 45 days visit compared with basal value
Adverse effects | Through study completion, an average of 9 months
  Any adverse effect (symptom, illness or other event of medical relevance) experienced by the participant during the course of the study or detected by the physician will be recorded in the data collection notebook, regardless of whether its nature may or may not be associated with the product in study. The registry of adverse effects will detail the nature of the adverse effect, its severity, the time of appearance and duration, the actions necessary for its treatment (if necessary) and the potential relationship with the treatment of the study, as well as any other relevant information .

SECONDARY OUTCOMES:
Concentration of S. mutans | Through study completion, an average of 9 months
  Concentration of S. mutans analysed by qPCR obtained from saliva and plaque samples at days 15, 30 and 45 compared with basal value
Concentration of S. dentisani | Through study completion, an average of 9 months
  Concentration of S. dentisani analysed by qPCR obtained from saliva and plaque samples at days 15, 30 and 45 compared with basal value
Lactic acid quantification before and after a sugar shock | Through study completion, an average of 9 months
  Quantification of lactic acid of the plaque ex vivo before and after a sugar shock measured in the RQflex 10 reflectometer by using Reflectoquant strips for lactate at days 15, 30 and 45 compared with basal value
pH quantification before and after a sugar shock | Through study completion, an average of 9 months
  Quantification of pH of the plaque ex vivo before and after a sugar shock measured in the RQflex 10 reflectometer by using Reflectoquant strips for pH at days 15, 30 and 45 compared with basal value
Salivary pH before and after a sugar shock | Through study completion, an average of 9 months
  Increase in salivary pH measured on the RQflex 10 reflectometer using Reflectoquant test strips at 15, 30 and 45 days visit compared with basal value after a sugar shock consisting in rinsing and active movements for 1 minute of a sterile 10% glucose solution.
Caries | Through study completion, an average of 9 months
  Occurrence of caries at 15, 30 and 45 days visit compared with basal value
Plaque | Through study completion, an average of 9 months
  Decrease in plaque index at 15, 30 and 45 days visit compared with basal value
Buffer capacity of the saliva | Through study completion, an average of 9 months
  Buffer capacity of the saliva measured by reactive strips, which determine the amount of acid that the saliva is capable of neutralizing at 15, 30 and 45 days visit compared with basal value

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Conde, Study Director — Effice
Locations (1):
- Lluis Alcanyis Foundation dental clinic, University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No